CLINICAL TRIAL: NCT02901028
Title: Safety Testing of an Innovative Concussion Prevention Device
Brief Title: Innovative Concussion Prevention Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013-2240
Record Dates: First submitted 2015-10-20; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collar Device (Experimental): The Device is a standard hockey neck guard, adapted for the purposes of this study. The Device incorporates two bulges localized over the site of the internal jugular veins bilaterally. Experiments performed with jugular Doppler ultrasound demonstrate that while wearing the Device, flows within the jugular veins are reduced, while flow within the carotid arteries and all portions of the cerebrum are preserved (JA Fisher, unpublished data). Thus, application of the Device to the subject will not cause any untoward health risks. The pressure exerted by the Device on the region of the neck superficial to the internal jugular vein is akin to the pressure felt when a person yawns or wears a snugly fitting necktie.
  Interventions: Other: Laboratory testing; Other: Blood and Urine Draws
- Arm Device (Sham Comparator): the subject is wearing a sham arm device, which will be placed on the upper arm and not cause venous engorgement. The subject will undergo the same testing as when wearing the collar device (strength, Vo2, vision, blood, urine, etc)
  Interventions: Other: Laboratory testing; Other: Blood and Urine Draws

INTERVENTIONS:
Other: Laboratory testing — Subjects will visit the Human Performance Laboratory on two separate occasions to perform the testing procedures. testing consists of VO2, strength, biomechanics, dynavision, etc.
Other: Blood and Urine Draws — subjects will have a blood draw and provide a urine sample

SUMMARY:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs currently being experienced for life-treatment of surviving victims. An externally-worn medical device that applies mild jugular compression according to the principle of the Queckenstedt Maneuver. PURPOSE: To monitor changes in vital signs, blood physiologies, oxygen consumption, biomechanics, strength, neurological capabilities, and balance in a population of athletes wearing the Device. Secondly, to determine the tolerance and acceptance of the Device while undergoing exertion.

DETAILED DESCRIPTION:
The Device has the promise of providing a novel mechanism for reducing or preventing the likelihood of TBI, and may be used in conjunction with other protective equipment. TBI is the leading cause of death in individuals under age 45. The cost of TBI in the U.S. is estimated at anywhere from $50 to $150 billion, annually. The January, 2008 New England Journal of Medicine reports, "Head and neck injuries, including severe brain trauma, have been reported in one quarter of service members who have been evacuated from Iraq and Afghanistan"[1-3]. The vast majority of these injuries have resulted from exposure to improvised explosive device (IED) blast waves. Head injuries, concussions and the resulting trauma have been in public discussion recently as the National Football League (NFL) deals with a lawsuit regarding head injuries by about one-third of living former NFL players and are also a concern for athletes who participate in a wide range of sports, including hockey, rugby and soccer.

According to NASA, "The oscillation of a fluid caused by external force, called sloshing, occurs in moving vehicles containing liquid masses, such as trucks, etc." This oscillation occurs when a vessel is only partially filled. Similarly, the brain faces slosh peril during external force impartation. Slosh permits external energies to be absorbed by the contents of a partially filled vessel or container by means of inelastic collisions. Tissues of differing densities can decelerate at different rates creating shear and cavitation. If the collisions between objects or molecules are elastic, the transfer of energies to those objects diminishes, minimizing the energies imparted by slosh.

Woodpeckers, head ramming sheep and all mammals (including mankind) have small, little known and misunderstood muscles in their necks called the omo-hyoid muscles. Highly G-tolerant creatures of the forest have utilized these muscles to gently restrict outflow of the internal jugular veins thereby "taking up" the excess compliance of the cranial space and ultimately protecting themselves from TBI like tiny "airbags" in a motor vehicle.

This study utilizes a randomized cross over study design. Subjects will visit the Human Performance Laboratory on two separate occasions to perform the testing procedures listed in the table below. During one testing session, the subject will perform the testing procedures while wearing the Device under investigation while the other testing session will be completed while the subject is wearing a sham arm device, which will be placed on the upper arm and not cause venous engorgement. The order of the testing sessions will be randomized prior to the subject's arrival for the first session. The Device is a standard hockey neck guard, adapted for the purposes of this study. The Device incorporates two bulges localized over the site of the internal jugular veins bilaterally. Experiments performed with jugular Doppler ultrasound demonstrate that while wearing the Device, flows within the jugular veins are reduced, while flow within the carotid arteries and all portions of the cerebrum are preserved (JA Fisher, unpublished data). Thus, application of the Device to the subject will not cause any untoward health risks. The pressure exerted by the Device on the region of the neck superficial to the internal jugular vein is akin to the pressure felt when a person yawns or wears a snugly fitting necktie.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Able to provide written consent
* Able to tolerate hypercapnia for 1-2 minutes
* Must be 18 years or older

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or head trauma
* Medical contraindications to limited hypercapnia or restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Known open eye injuries
* Neck injuries
* Any known airway obstruction
* Any known seizure disorder
* Any altered level of consciousness
* Have suffered an injury to a lower extremity in the past 6 months
* Have undergone ACL reconstruction less than 2 years ago
* Cardiovascular/Respiratory issues

  * Known untreated hypertension
  * Known cardiomyopathy
  * Known exercise intolerance
* Any indication of cardiovascular risk by the Physical Activity Readiness Questionnaire (PAR-Q)
* Under the age of 18 years

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Measure any changes in blood physiologies | 1 week
  To monitor changes blood physiologies in a population of athletes wearing the Device.
measure any changes in oxygen consumption | 1 week
  To monitor changes oxygen consumption in a population of athletes wearing the Device.
measure any changes in strength | 1 week
  To monitor changes in strength in a population of athletes wearing the Device.
Measure any changes in biomechanics | 1 week
  To monitor changes in biomechanics balance in a population of athletes wearing the Device.
Measure any changes in neurological capabilities | 1 week
  To monitor changes in neurological capabilities in a population of athletes wearing the Device.
Measure any changes in balance | 1 week
  To monitor changes in and balance in a population of athletes wearing the Device.

SECONDARY OUTCOMES:
Number of participants with intervention-related adverse events as assessed by participant survey | 1 week
  to determine the tolerance and acceptance of the Device while undergoing exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published however individual participant data will remain secure